CLINICAL TRIAL: NCT03635749
Title: Intensive Statin and Antiplatelet Therapy for High-risk Intracranial or Extracranial Atherosclerosis (INSPIRES)
Brief Title: Intensive Medical Therapy for High-risk Intracranial or Extracranial Atherosclerosis
Acronym: INSPIRES
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017YFC1307905
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Acute Stroke; Transient Ischemic Attack
Keywords: Acute Stroke; Transient Ischemic Attack; Antiplatelet Therapy; Randomized Controlled Trial; Double Blind Study; Multicenter Study; Symptomatic Extracranial or Intracranial Arterial Stenosis; Statin Therapy; Clinical Trial
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: The subjects are randomly assigned to the following four groups:
  1. Intensive antiplatelet therapy + immediate high-intensity statin therapy (80mg atorvastatin)
  2. Intensive antiplatelet therapy + delayed high-intensity statin therapy (40mg atorvastatin)
  3. Standard antiplatelet therapy + immediate high-intensity statin therapy (80mg atorvastatin)
  4. Standard antiplatelet therapy + delayed high-intensity statin therapy (40mg atorvastatin)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two nearly identical tablet forms of Clopidogrel (75mg Clopidogrel and matching placebo) with almost the same size, color and smell will be used in this research.
  Two nearly identical tablet forms of Aspirin (100mg Aspirin and matching placebo) with almost the same size, color and smell will be used in this research.
  Two nearly identical tablet forms of Atorvastatin (20mg Atorvastatin and matching placebo) with almost the same size, color and smell will be used in this research.
  Centers are not able to apply unblinding with biological experiment in this study. Researchers shall never unblind the code unless special situations occur such as Serious Adverse Events (SAE), which is essential for treatment. Clinical outcomes of efficacy and safety are submitted to Adjudication Committee, who should be blinded to randomization, for final determination.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DAPT + immediate high-intensity statin (Active Comparator): This group will receive active clopidogrel and active aspirin (Dual antiplatelet therapy, DAPT); active atorvastatin calcium with high dosage in the early phase.
  Interventions: Drug: Intensive antiplatelet; Drug: Immediate high-intensity statin
- DAPT + delayed high-intensity statin (Other): This group will receive active clopidogrel and active aspirin (Dual antiplatelet therapy, DAPT); atorvastatin calcium placebo and active atorvastatin calcium with moderate dosage in the ealy phase.
  Interventions: Drug: Intensive antiplatelet; Drug: Delayed high-intensity statin
- Aspirin+immediate high-intensity statin (Other): This group will receive active aspirin and clopidogrel placebo; active atorvastatin calcium with high dosage in the early phase.
  Interventions: Drug: Standard antiplatelet; Drug: Immediate high-intensity statin
- Aspirin+delayed high-intensity statin (Placebo Comparator): This group will receive active aspirin and clopidogrel placebo; atorvastatin calcium placebo and active atorvastatin calcium with moderate dosage in the early phase.
  Interventions: Drug: Standard antiplatelet; Drug: Delayed high-intensity statin

INTERVENTIONS:
Drug: Intensive antiplatelet — Day 1：clopidogrel 300mg/day+ aspirin100-300mg/ day
  Day2 - 21: clopidogrel 75mg/day+ aspirin 100mg/day
  Day22 - 90: clopidogrel 75mg/day+aspirin placebo
  Other Names: Dual antiplatelet
  Arms: DAPT + delayed high-intensity statin; DAPT + immediate high-intensity statin
Drug: Standard antiplatelet — Day 1: Aspirin 100-300mg/day + clopidogrel placebo
  Day 2 - 90: Aspirin 100mg/day+ clopidogrel placebo
  Other Names: Aspirin
  Arms: Aspirin+delayed high-intensity statin; Aspirin+immediate high-intensity statin
Drug: Immediate high-intensity statin — Day 1 - 21：Atorvastatin calcium 80mg/day
  Day 22 - 90：Atorvastatin calcium 40mg/day
  Other Names: Immediate Atorvastatin
  Arms: Aspirin+immediate high-intensity statin; DAPT + immediate high-intensity statin
Drug: Delayed high-intensity statin — Day 1 - 3：Atorvastatin calcium placebo
  Day 4 - 21：Atorvastatin calcium 40mg/day + Atorvastatin calcium placebo
  Day 22 - 90：Atorvastatin calcium 40mg/day
  Other Names: Delayed Atorvastatin
  Arms: Aspirin+delayed high-intensity statin; DAPT + delayed high-intensity statin

SUMMARY:
Large-artery stenosis plays an important role in the occurrence of ischemic stroke. The primary purpose of this study is to evaluate the efficacy and safety of intensive antiplatelet therapy versus standard antiplatelet therapy and immediate high-intensity statin therapy (80mg atorvastatin) versus delayed high-intensity statin therapy (40mg atorvastatin) and intensive antiplatelet combined with immediate high-intensity statin therapy (80mg atorvastatin) versus standard antiplatelet combined with delayed high-intensity statin therapy (40mg atorvastatin) in reducing the risk of stroke at 90 days in patients with acute and high-risk symptomatic extracranial or intracranial arterial stenosis.

DETAILED DESCRIPTION:
Large-artery atherosclerotic stenosis is the main cause of ischemic stroke, especially in Asian population. However, targeted treatment evidence for large-artery atherosclerotic stenosis is limited according to the current guidelines. And also, randomized trial for statin therapy in patients with acute large arterial stenosis at early stage is still limited. The primary purpose of this study is to evaluate the efficacy and safety of intensive antiplatelet therapy versus standard antiplatelet therapy in reducing the risk of stroke at 90 days in patients with acute and high-risk symptomatic extracranial or intracranial arterial stenosis; the efficacy and safety of immediate high-intensity statin therapy (80mg atorvastatin) versus delayed high-intensity statin therapy (40mg atorvastatin) in reducing the risk of stroke at 90 days in patients with acute and high-risk symptomatic extracranial or intracranial arterial stenosis; and the efficacy and safety of intensive antiplatelet combined with immediate high-intensity statin therapy (80mg atorvastatin) versus standard antiplatelet combined with delayed high-intensity statin therapy (40mg atorvastatin) in reducing the risk of stroke at 90 days in patients with acute and high-risk symptomatic extracranial or intracranial arterial stenosis.

This trial is a randomized, double-blind, placebo-controlled, multicenter, 2×2 factorial designed clinical trial. 6100 patients in 250 centers in China will be enrolled with one of the following situations (1) Mild ischemic stroke (NIHSS 4~5) within 24 hours of onset meets any of the following imaging conditions: a) Acute single cerebral infarction with criminal intracranial and extracranial atherosclerotic stenosis (stenosis rate ≥50%),b) Acute multiple cerebral infarction (considered to be caused by large artery atherosclerosis, including non-stenotic vulnerable plaque);Or (2) Moderate-to-high-risk TIA (ABCD2≥4) or mild ischemic stroke (NIHSS≤5) within 24 to 72 hours of onset meets any of the following imaging conditions: a) Medium and high risk TIA with criminal intracranial and extracranial atherosclerotic stenosis (stenosis rate ≥50%),b) Acute single cerebral infarction with criminal intracranial and extracranial atherosclerotic stenosis (stenosis rate ≥50%),c) Acute multiple cerebral infarction (considered to be caused by large artery atherosclerosis, including non-stenotic vulnerable plaque) . Patients will be randomly assigned into 4 groups according to the ratio of 1:1:1:1:

1. Intensive antiplatelet therapy + immediate high-intensity statin therapy (80mg atorvastatin)
2. Intensive antiplatelet therapy + delayed high-intensity statin therapy (40mg atorvastatin)
3. Standard antiplatelet therapy + immediate high-intensity statin therapy (80mg atorvastatin)
4. Standard antiplatelet therapy + delayed high-intensity statin therapy (40mg atorvastatin)

Face to face interviews will be made at baseline, 7, 14 (or hospital discharge), 90 ± 7 days and 12th month ± 14 days after randomization.

Survival curves will be estimated for the primary outcome using the Kaplan-Meier procedure and compared using a Cox regression model Wald test, stratified by the opposite arm of the factorial design. Safety outcomes will be calculated using the Kaplan-Meier curve to simulate the 3-month cumulative risk, and the Cox proportional hazards model to calculate the HR and 95% confidence interval.

Primary outcome is defined as stroke (including hemorrhagic and ischemic stroke). Secondary outcomes include composite vascular events (stroke, myocardial infarction, and cardiovascular death); ischemic stroke; transient ischemic attack; myocardial infarction; vascular death; all-cause death; poor functional outcome (mRS 2-6); and quality of life (EQ-5D scale). Safety outcomes, relating to antiplatelet therapy (i.e. bleeding, intracranial hemorrhage, and adverse events) and statin therapy (i.e. hepatotoxicity, muscle toxicity and adverse events) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Age :35-80 years old , male or female;
2. Any of the following three two situations:

(1) Mild ischemic stroke (NIHSS 4 to 5 points) within 24 hours of onset meets any of the following imaging conditions:

1. Acute single cerebral infarction with criminal intracranial and extracranial atherosclerotic stenosis (stenosis rate ≥50%)
2. Acute multiple cerebral infarction (considered to be caused by large artery atherosclerosis, including non-stenotic vulnerable plaque)

Or (2) Moderate-to-high-risk TIA (ABCD2≥4 points) or mild ischemic stroke (NIHSS≤5 points) within 24 to 72 hours of onset meets any of the following imaging conditions:

1. Medium and high risk TIA with criminal intracranial and extracranial atherosclerotic stenosis (stenosis rate ≥50%)
2. Acute single cerebral infarction with criminal intracranial and extracranial atherosclerotic stenosis (stenosis rate ≥50%)
3. Acute multiple cerebral infarction (considered to be caused by large artery atherosclerosis, including non-stenotic vulnerable plaque)

The rate of intracranial artery stenosis is assessed by MRA, CTA, or DSA according to WASID standards; the rate of extracranial artery stenosis is assessed by carotid ultrasound, CEMRA, CTA or DSA, according to NASCET standards; 3. Signed informed consent

Exclusion Criteria:

1. Specific cardiogenic ischemic cerebrovascular diseases(eg. combined with atrial fibrillation, heart valve prosthesis, atrial myxoma, endocarditis, etc.)
2. Other ischemic cerebrovascular diseases with specific causes (eg. aortic dissection, vasculitis, vascular malformation, etc.)
3. Non-cerebral vascular disease (eg. intracranial tumors, multiple sclerosis)
4. Cerebral infarction of large area (infarct size greater than half the single lobe area)
5. CT indicating hemorrhagic transformation of cerebral infarction before randomization
6. Patients with pre-existing contraindications of using clopidogrel, aspirin or statin drugs:

   Known history of allergy ; Severe heart failure and asthma ; Coagulant disorders and systemic bleeding ; Pre-existing drug - induced blood system disease or abnormal liver function ; Leukopenia (< 2×109/l) or thrombocytopenia (<100×109/l) ; active liver disease ; pregnancy or lactation period ; Severe heart failure：New York Heart Association (NYHA) Functional Classification III and IV
7. MRS > 2 before the onset
8. Use of intravenous or arterial thrombolysis intravascular therapy or bridge therapy after onset
9. Use of defibrinating therapy like snake venom, defibrase, lumbrokinase, etc. or use of anticoagulant therapy like argatroban, or use of antiplatelet therapy except clopidogrel and aspirin, such as tirofiban, ticagrelor, ozagrel, and so on after onset.
10. Creatine Kinase(CK) more than 5 times of the upper limit of normal value after onset
11. Use of drugs affecting the metabolism of statins such as immune-suppressive drugs, antifungal agents, or fibrates drugs and so on, within 14 days before randomization.
12. Severe hepatic or renal insufficiency (Note: Severe hepatic insufficiency refers to the ALT value > 2 times the upper limit of normal value or AST times > 2 times the upper limit of normal value; Severe hepatic insufficiency is refers to creatinine values > 1.5 times he upper limit of normal value or GFR < 40 ml/min/1.73 m2)
13. Usage of dual antiplatelet therapy with aspirin plus clopidogrel within 14 days before randomization. (patients who received dual antiplatelet therapy (aspirin combined with clopidogrel) but did not use clopidogrel with loading dose after onset were excluded)
14. Use of Intensive statin therapy within 14 days before randomization（atorvastatin ≥40mg/d or rosuvastatin ≥ 20mg/d）.
15. Pre-existing intracranial hemorrhage（eg. ICH, SAH）
16. Gastrointestinal bleeding or major surgery occurred within 90 days before randomization.
17. Pre-existing extracranial angioplasty or vascular surgery
18. Anticipated requirement for long-term non-study antiplatelet drugs, or non-steroid anti-inflammatory drugs.
19. Experimental drugs need to stop due to angioplasty or vascular surgery, which was planned or likely to perform within 90 days after randomization
20. Patients with severe disease expected to live for less than 90 days
21. Pregnant or childbearing-age women who have no effective contraceptives or positive pregnancy test records
22. Patients who are undergoing experimental drugs or device tests
23. Unable to finish the follow-up of 90 days due to geographical factor or other reasons（eg. dementia, alcoholism, substance abuse, severe mental disease, etc.）

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6100 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Stroke | 90 days
  Symptoms and signs of acute neurological deficits caused by sudden focal or whole brain, spinal cord or retinal vascular damage, which are related to cerebral circulatory disorders, including hemorrhagic and ischemic stroke

SECONDARY OUTCOMES:
Composite vascular events | 90 days
  stroke (including hemorrhagic and ischemic stroke), myocardial infarction, and cardiovascular death.
Ischemic stroke | 90 days
  An acute focal infarction of the brain or retina. Criteria:(1) acute onset of a new focal neurological deficit with clinical or imaging evidence of infarction lasting more than 24 hours and not attributable to a non-ischemic etiology (not associated with brain infection, trauma, tumor, seizure, severe metabolic disease, or degenerative neurological disease); or (2) acute onset of a new focal neurological deficit and not attributable to a non-ischemic etiology lasting less than 24 hours, but accompanied by neuroimaging evidence of new brain infarction; or, (3) rapid worsening of an existing focal neurological deficit (an increase in NIHSS of ≥4 on the basis of a primary ischemic stroke, excluding hemorrhagic transformation or symptomatic cranial disease after infarction) lasting more than 24 hours and not attributable to a non-ischemic etiology, and accompanied by new ischemic changes on brain MRI or CT.
Transient ischemic attack | 90 days
  A neurological deficit of sudden onset, resolving completely, attributed to focal brain or retinal ischemia without evidence of associated acute focal infarction of the brain. Criteria: rapid onset of a focal neurological deficit that is without evidence of acute focal infarction of the brain, and is not attributable to a non-ischemic etiology (brain infection, trauma, tumor, seizure, severe metabolic disease, or degenerative neurological disease)
Myocardial infarction | 90 days
  Acute myocardial infarction is diagnosed by the third edition of the international general diagnostic criteria (Glob Heart. 2012 Dec;7(4):275-95)
Vascular death | 90 days
  Vascular death includes stroke, sudden cardiac death, acute myocardial infarction, heart failure, pulmonary embolism, heart / cerebrovascular intervention or surgery (death unrelated to acute MI) and other cardiovascular causes of death [such as: Arrhythmia irrelevant with sudden cardiac death, aortic aneurysm rupture, or peripheral artery disease. Any death of unknown/unclear cause that occurs within 30 days after stroke, myocardial infarction, or cardio-cerebrovascular operation/surgery will be regarded as death due to stroke, myocardial infarction, or cardio-cerebrovascular operation/surgery, respectively.
All-cause death | 90 days
  All-cause death
Poor functional outcome | 90 days
  The modified Rankin Scale (mRS)= 2-6
Quality of life (EQ-5D scale) | 90 days
  EQ-5D scale index score ≤0.5
Change of atherosclerotic plaque using high-resolution magnetic resonance imaging (HR-MRI) | 90 days
  Change of atherosclerotic plaque using high-resolution magnetic resonance 。 Patients in HR-MRI subgroup only
Early Neurological Deficits | 7 days
  NIHSS score increase of no less than 2points
Ordinal stroke or TIA | 90 days
  The new stroke or TIA is classified on a six-level ordered category scale combined vascular events with mRS score at 90 days or at 1year, respectively: fatal stroke (stroke with subsequent death), severe stroke (stroke followed by mRS of 4-5), moderate stroke (stroke followed by mRS of 2-3), mild stroke (stroke followed by mRS of 0-1), TIA and no stroke/TIA.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, MD, PhD, Principal Investigator — Beijing Tiantan Hospital
Locations (113):
- China (113):
  - Tiantan Hospital, Beijing, Beijing Municipality
  - Anshan Central Hospital, Anshan
  - General Hospital of Anshan Iron and Steel Company, Anshan
  - Anyang People's Hospital, Anyang
  - Baoding First Central Hospital, Baoding
  - Beijing Hepingli Hospital, Beijing
  - Benxi Central Hospital, Benxi
  - First Hospital of Changsha, Changsha
  - Second people's Hospital of Hunan Province, Changsha
  - Xiangya Third Hospital of Central South University, Changsha
  - Changzhi Medical College Affiliated Heping Hospital, Changzhi
  - Changzhi People's Hospital, Changzhi
  - Lu'an Group General Hospital, Changzhi
  - Changzhou Second People's Hospital, Changzhou
  - Changzhou Wujin Hospital of Traditional Chinese Medicine, Changzhou
  - Chongqing Sanxia Central Hospital, Chongqing
  - Southwest Hospital affiliated to the Army Military Medical University, Chongqing
  - People's Hospital of Dali Bai Autonomous Prefecture, Dali
  - Dalian Central Hospital, Dalian
  - Dalian Friendship Hospital, Dalian
  - Second people's Hospital of Dalian, Dalian
  - Xinhua Hospital Affiliated to Dalian University, Dalian
  - Datong Third People's Hospital, Datong
  - Dazhou Central Hospital, Dazhou
  - Dongguan Hong Wah hospital, Dongguan
  - Donghua Hospital, Dongguan
  - Dongyang People's Hospital, Dongyang
  - People's Hospital of Dongying District, Dongying
  - General Hospital of Fushun Mining Bureau, Fushun
  - Fuxin Mining Group General Hospital, Fuxin
  - Nanxi Mountain hospital in Guangxi District, Guilin
  - Guiyang Second Hospital, Guiyang
  - Handan Central Hospital, Handan
  - Handan First Hospital, Handan
  - General Hospital of the General Administration of agriculture and reclamation of Heilongjiang, Ha’erbin
  - Second hospital of Hebei Medical University, Hebei
  - Hengshui Sixth People's Hospital, Hengshui
  - Nanhua Hospital Affiliated to Nanhua University, Hengyang
  - The Inner Mongolia Autonomous Region people's Hospital, Hohhot
  - First Affiliated Hospital of Jiamusi University, Jiamusi
  - Jiamusi Central Hospital, Jiamusi
  - Jilin Electric Power Hospital, Jilin
  - Jinlin Central Hospital, Jilin
  - Jinlin People's Hospital, Jilin
  - Second hospital of Jilin University, Jilin
  - Qianfo Hill Hospital of Shandong Province, Jinan
  - Shandong Transportation Hospital, Jinan
  - Affiliated Hospital of Jiujiang University, Jiujiang
  - Jixi People's Hospital, Jixi
  - Kaifeng Central Hospital, Kaifeng
  - Liaocheng Brain Hospital, Liaocheng
  - Liaocheng Second People's Hospital, Liaocheng
  - Liaoyang Central Hospital, Liaoyang
  - Linfen People's Hospital, Linfen
  - Second Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Luzhou Hospital of traditional Chinese Medicine, Luzhou
  - Mishan People's Hospital, Mishan
  - Mudanjiang Second People's Hospital, Mudanjiang
  - Fourth Affiliated Hospital of Nanchang University, Nanchang
  - Third Affiliated Hospital of Nanchang University, Nanchang
  - Wuxi Affiliated Hospital of Nanjing University of Chinese Medicine, Nanjing
  - Li Huili Hospital of Ningbo Medical Center, Ningbo
  - Ningbo Second Hospital, Ningbo
  - Ningde People's Hospital, Ningde
  - Panjin Central Hospital, Panjin
  - Pindingshan First People's Hospital, Pingdingshan
  - Qiqihar First Hospital, Qiqihar
  - Ruzhou First People's Hospital, Rizhao
  - Sanmenxia Central Hospital, Sanmenxia
  - Fifth People's Hospital of Shanghai City, affiliated to Fudan University, Shanghai
  - Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai
  - Second hospital of Shanxi Medical University, Shanxi
  - Shengzhou People's Hospital, Shaoxing
  - Heilongjiang Agriculture and Reclamation Bei'an Administration Central Hospital, Shenyang
  - Shenzhen Second People's Hospital, Shenzhen
  - Shijiazhuang Pingan Hospital, Shijiazhuang
  - First Hospital Affiliated to Suzhou University, Suzhou
  - The Second Hospital Affiliated to Suzhou University, Suzhou
  - Taizhou First People's Hospital, Taizhou
  - Affiliated Hospital of North China Polytechnic University, Tangshan
  - Tangshan Workers' Hospital, Tangshan
  - Tianjin Fourth Central Hospital, Tianjin
  - Tieling Central Hospital, Tieling
  - Gaomi People's Hospital, Weifang
  - People's Hospital of Wendeng District, Weihai
  - People's Hospital of Wuhan University, Wuhan
  - Wuhan Central Hospital, Wuhan
  - Gansu Academy of Medical Sciences, Wuwei, Wuwei
  - Wuxi People's Hospital, Wuxi
  - Wuxi Second People's Hospital, Wuxi
  - Xi'an 141 hospital, Xi'an
  - Xian First Hospital, Xi'an
  - Xinxiang Central Hospital, Xinxiang
  - Xinyang Central Hospital, Xinyang
  - Xuchang Central Hospital, Xuchang
  - General Hospital of Xuzhou Mining Group, Xuzhou
  - Xuzhou First People's Hospital, Xuzhou
  - Yantai Yuhuangding Hospital Affiliated to Qiingdao University, Yantai
  - Yibin First People's Hospital, Yibin
  - Yichang First People's Hospital, Yichang
  - Yingkou Central Hospital, Yingkou
  - Yueyang Hospital of integrated traditional Chinese and Western Medicine Affiliated to Shanghai University of Traditional Chinese Medicine, Yueyang
  - Dehong People's Hospital of Yunnan, Yunnan
  - Zaozhuang Mining Group Zaozhuang hospital, Zaozhuang
  - Zhangjiagang First People's Hospital, Zhangjiagang
  - Zhangjiagang Traditional Chinese Medicine Hospital, Zhangjiagang
  - Workers' Hospital of Hebei iron and Steel Group Xuanhua iron and Steel Co., Ltd., Zhangjiakou
  - Central Hospital of the Yellow River, Zhengzhou
  - Zhengzhou First People's Hospital, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang
  - Zhoukou Yongshan hospital, Zhoukou
  - Zhumadian Central Hospital, Zhumadian
  - Zigong First People's Hospital, Zigong

REFERENCES:
- [Derived] Liu C, Li Y, Liu Z, Gao Y, Zhang Q, Wabnitz AM, Pan Y, Yan H, Chen W, Johnston SC, Wang D, Amarenco P, Bath PM, Wang Y, Wang Y, Guan L. The effect of dual antiplatelet therapy in different patterns of watershed infarction: Subgroup analysis of the INSPIRES trial. Cell Rep Med. 2026 Feb 5:102596. doi: 10.1016/j.xcrm.2026.102596. Online ahead of print. PMID 41650951
- [Derived] Chen Y, Jiang L, Gao Y, Chen W, Yan H, Wang T, Yang Y, Yao D, Liu D, Pan Y, Wang Y. CYP2C19 Genotype and Efficacy of Clopidogrel Initiated Between 24 to 72 Hours for Ischemic Stroke. Stroke. 2025 Nov;56(11):3108-3117. doi: 10.1161/STROKEAHA.125.052167. Epub 2025 Sep 18. PMID 40964718
- [Derived] Xia Z, Gao Y, Chen W, Johnston SC, Amarenco P, Bath PM, Wang X, Yan H, Wang T, Yang Y, Zhang Y, Wang M, Jing J, Wang C, Wang Y, Wang Y, Pan Y. Dual Antiplatelet Therapy in Patients With Metabolic Syndrome After Mild Ischemic Stroke or Transient Ischemic Attack. J Am Heart Assoc. 2025 Aug 5;14(15):e041449. doi: 10.1161/JAHA.125.041449. Epub 2025 Jul 17. PMID 40673545
- [Derived] Liu D, Yan H, Gao Y, Chen W, Johnston SC, Amarenco P, Bath PM, Wang X, Wang M, Wang T, Yang Y, Jing J, Wang C, Wang Y, Pan Y, Wang Y. Effect of history of hypertension on efficacy of clopidogrel-aspirin in ischemic stroke. Int J Stroke. 2025 Oct;20(8):1021-1030. doi: 10.1177/17474930251338618. Epub 2025 Apr 19. PMID 40251953
- [Derived] Li H, Cheng M, Gao Y, Yan H, Wang Y, Johnston SC, Bath PM, Amarenco P, Yang Y, Chen W, Wang Y, Pan Y, Wang Y. Does the Burden of CSVD Modify the Efficacy of Dual Antiplatelet Therapy?: A Post Hoc Analysis of the INSPIRES Trial. Stroke. 2025 Jun;56(6):1376-1387. doi: 10.1161/STROKEAHA.124.049826. Epub 2025 Apr 7. PMID 40190261
- [Derived] Zhou Q, Gao Y, Chen W, Johnston SC, Amarenco P, Bath PM, Wang X, Yan H, Wang T, Yang Y, Zhang Y, Yang Q, Wang M, Jing J, Wang C, Wang Y, Wang Y, Pan Y. Efficacy and Safety of Dual Antiplatelet Treatment up to 72 Hours in Acute Ischemic Stroke Stratified by Glycemic Status. Ann Neurol. 2025 Jul;98(1):174-182. doi: 10.1002/ana.27207. Epub 2025 Feb 11. PMID 39931900
- [Derived] Zhang Y, Wang X, Gao Y, Chen W, Johnston SC, Amarenco P, Bath PM, Yan H, Wang T, Yang Y, Zhou Q, Wang M, Jing J, Wang C, Wang Y, Wang Y, Pan Y. Dual Antiplatelet Treatment up to 72 Hours After Ischemic Stroke Stratified by Risk Profile: A Post Hoc Analysis. Stroke. 2025 Jan;56(1):46-55. doi: 10.1161/STROKEAHA.124.049246. Epub 2024 Dec 20. PMID 39705390
- [Derived] Guan L, Han S, Johnston SC, Bath PM, Amarenco P, Yang Y, Wang T, Jing J, Wang C, Gao Y, Chen W, Yan H, Wang X, Wang Y, Wang Y, Pan Y. Duration of Benefit and Risk of Dual Antiplatelet Therapy up to 72 Hours After Mild Ischemic Stroke and Transient Ischemic Attack. Neurology. 2024 Oct 8;103(7):e209845. doi: 10.1212/WNL.0000000000209845. Epub 2024 Sep 13. PMID 39270151
- [Derived] Liu Y, Zhao J, Gao Y, Chen W, Johnston SC, Bath PM, Amarenco P, Yan H, Wang X, Yang Y, Wang T, Wang Y, Pan Y, Wang Y. Clopidogrel and Aspirin Initiated Between 24 to 72 Hours for Mild Ischemic Stroke: A Subgroup Analysis of the INSPIRES Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2431938. doi: 10.1001/jamanetworkopen.2024.31938. PMID 39240565
- [Derived] Gao Y, Jiang L, Pan Y, Chen W, Jing J, Wang C, Johnston SC, Amarenco P, Bath PM, Yang Y, Wang T, Han S, Meng X, Lin J, Zhao X, Liu L, Zhao J, Li Y, Zang Y, Zhang S, Yang H, Yang J, Wang Y, Li D, Wang Y, Liu D, Kang G, Wang Y, Wang Y; INSPIRES Investigators. Immediate- or Delayed-Intensive Statin in Acute Cerebral Ischemia: The INSPIRES Randomized Clinical Trial. JAMA Neurol. 2024 Jul 1;81(7):741-751. doi: 10.1001/jamaneurol.2024.1433. PMID 38805216
- [Derived] Gao Y, Chen W, Pan Y, Jing J, Wang C, Johnston SC, Amarenco P, Bath PM, Jiang L, Yang Y, Wang T, Han S, Meng X, Lin J, Zhao X, Liu L, Zhao J, Li Y, Zang Y, Zhang S, Yang H, Yang J, Wang Y, Li D, Wang Y, Liu D, Kang G, Wang Y, Wang Y; INSPIRES Investigators. Dual Antiplatelet Treatment up to 72 Hours after Ischemic Stroke. N Engl J Med. 2023 Dec 28;389(26):2413-2424. doi: 10.1056/NEJMoa2309137. PMID 38157499
- [Derived] Gao Y, Pan Y, Han S, Chen W, Jing J, Wang C, Yang Y, Wang T, Meng X, Zhao X, Liu L, Li H, Johnston SC, Amarenco P, Bath PM, Wang Y, Wang Y; INSPIRES Investigators. Rationale and design of a randomised double-blind 2x2 factorial trial comparing the effect of a 3-month intensive statin and antiplatelet therapy for patients with acute mild ischaemic stroke or high-risk TIA with intracranial or extracranial atherosclerosis (INSPIRES). Stroke Vasc Neurol. 2023 Jun;8(3):249-258. doi: 10.1136/svn-2022-002084. Epub 2023 Jan 27. PMID 36707080